CLINICAL TRIAL: NCT00469690
Title: Aqueous Concentrations and PGE2 Inhibition of Ketorolac 0.4% vs. Bromfenac 0.09% in Cataract Patients: Trough Drug Effects
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Innovative Medical (Industry)
Responsible Party: Frank Bucci, MD, Bucci Laser Vision Institute and Ambulatory Surgery Cneter
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 5305
Record Dates: First submitted 2007-05-02; First posted 2007-05-04 (Estimated); Last update posted 2008-05-20 (Estimated); Status verified 2008-05

CONDITIONS: Cataract
MeSH Terms: conditions — Cataract | interventions — Ketorolac Tromethamine; bromfenac

STUDY DESIGN:
Who Masked: Investigator

ARMS (2):
- 1 (Other)
  Interventions: Drug: Acular, Xibrom
- 2 (Other)
  Interventions: Drug: Acular, Xibrom

INTERVENTIONS:
Drug: Acular, Xibrom — 1. Acular 5ml (in the eye)Instill one drop into the eye to be operated on four times a day at (6am, 12pm, 6pm, 12am)
  2. Xibrom 5ml (in the eye) Instill one drop into the eye to be operated on two times a day (8am and 8pm)

SUMMARY:
The purpose of this study is to compare the ability of two different topical NSAIDs (non-steroidal anti-inflammatory medications used for pain relief) to reach the back of the eye and to stop inflammation. The study will conclude on the day of your cataract surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy Male/Female 21 years of age of older.
2. Patient understands and is willing to sign the written informed consent form
3. Likely to complete the entire course of the study.
4. Patient is scheduled to undergo cataract surgery
5. Female patients of childbearing potential must have had a regular menstrual cycle prior to study entry (a female is considered of childbearing potential unless she is postmenopausal, without a uterus and/or both ovaries, or has had a bilateral tubal ligation).
6. Patient is willing and able to administer eye drops and record the times the drops were instilled

Exclusion Criteria:

1. Patient has been using a topical NSAID within 1 week of study entry
2. Patient has a known sensitivity to any of the ingredients in the study medications
3. Patient has sight in only one eye
4. Patient has a history of previous intraocular surgery
5. Patient's doctor has determined they have a condition (i.e., UNCONTROLLED systemic disease) or are in a situation that may put them at significant risk, confound the study results or may interfere significantly with their participation in the study
6. Female patients who are pregnant, nursing an infant or planning a pregnancy
7. Patients who are currently involved in another investigational study or have participated in one within the 30 days prior to entering this study

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2007-05; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
Aqueous concentrations | 8 months

SECONDARY OUTCOMES:
PGE2 Inhibition | 8 months

CONTACTS AND LOCATIONS:
Overall Officials: Frank Bucci, MD, Principal Investigator — Bucci Laser Vision Institute and Ambulatory Surgery Center
Locations (1):
- Bucci Laser Vision Institute and Ambulatory Surgery Center, Wilkes-Barre, Pennsylvania, United States